CLINICAL TRIAL: NCT00592410
Title: The Effects of Intensive Insulin on Somatic and Visceral Protein Turnover in Acute Kidney Injury (AKI)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Alp Ikizler, MD, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 061022
Record Dates: First submitted 2007-12-18; First posted 2008-01-14 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-08

CONDITIONS: Acute Renal Failure
MeSH Terms: conditions — Acute Kidney Injury | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: human regular insulin

INTERVENTIONS:
Drug: human regular insulin — administration of a primed continuous infusion of human regular insulin at a rate of 2.0 mU/kg/min while maintaining the plasma glucose level at 100 mg/dl via adjusting a variable infusion of 50% dextrose (i.e., a hyperinsulinemic euglycemic blood glucose clamp); duration of 3 hours; performed concomitantly with amino acid supplementation

SUMMARY:
We propose to determine the acute metabolic effects of intensive insulin therapy when administered to AKI patients with a particular focus on its effects on protein metabolism. We hypothesize that the degree of insulin resistance correlates with protein catabolism in critically ill patients with AKI, and that intensive insulin therapy will result in substantial reductions in both whole-body and skeletal muscle protein breakdown thereby improving overall protein balance. We also hypothesize that this therapy will have favorable effects on the inflammatory and oxidative stress profile of patients with AKI. The metabolic response to these interventions will be assessed through stable isotope infusion techniques, allowing for the most precise assessment of protein and energy homeostasis.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age admitted to the intensive care unit
* New onset acute kidney injury (AKI) or AKI superimposed on chronic kidney disease. AKI will be defined as:

  * an abrupt (within 48 hours) sustained increase (>24 hours) in serum creatinine of 2X baseline or
  * a reduction in urine output (documented oliguria of < 0.5 ml/kg/hr for >12 hours)
* Patients will be recruited for the study within 3-5 days following establishment of AKI

Exclusion Criteria:

* Institutionalized patient
* Unable to obtain consent from subject or legally recognized representative
* Pregnancy
* Patients receiving insulin within 12 hours of the study or patients with known diabetes mellitus.
* Patients receiving immunosuppressive medication including steroids (prednisone or equivalent dose ≥ 5 mg PO QD)
* AKI from urinary tract obstruction or a volume responsive pre-renal state.
* Liver Failure, defined as transaminase levels 3 times above the limit of normal or a total Bilirubin greater than 4 mg/dl.
* Evidence of active bleeding, defined as admission for bleeding (ex. GI bleed, ruptured aneurysm, trauma-related) coupled with an explained or unexplained decrease in hemoglobin of >2 points in the past 24 hours, or Hgb<8/Hct<24
* Ongoing myocardial ischemia or heart failure
* Life expectancy < 48 hours
* Patients without existing central venous access
* Hemodynamically unstable patients requiring active pressor titration, defined as an increase in current pressor dose by >20% or addition of a new pressor within 12 hours of initiating the study.
* History of Phenylketonuria (PKU) or other documented inborn errors of metabolism
* Hypokalemia, defined as a serum potassium of <3.0 mg/dl.
* Uncontrolled seizure disorder, defined as having seizure as a reason for admission, ongoing delirium tremens, or having had a seizure within 1 month of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
A change in whole body and muscle protein breakdown during amino acid supplementation with insulin versus baseline | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center